CLINICAL TRIAL: NCT04230473
Title: A Clinical Trial of CNCT19 Cells in the Treatment of CD19 Positive Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY-CD19 CART-001
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Relapsed or Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of CNCT19 (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CNCT19.
  Interventions: Biological: single dose of CNCT19

INTERVENTIONS:
Biological: single dose of CNCT19 — Dose A: 0.25 x 10^8 autologous CNCT19 transduced cells via intravenous infusion. Drug: Fludarabine Drug: Cyclophosphamide
  Dose B: 1.00 x 10^8 autologous CNCT19 transduced cells via intravenous infusion. Drug: Fludarabine Drug: Cyclophosphamide
  Dose C: 2.00 x 10^8 autologous CNCT19 transduced cells via intravenous infusion. Drug: Fludarabine Drug: Cyclophosphamide

SUMMARY:
This is a single arm, open-label, non-randomized, dose-escalation, phase I study to determine the safety and efficacy of CNCT19 in adult patients with relapsed or refractory acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
This is a single arm, open-label, non-randomized, dose-escalation, phase I study to determine the safety and efficacy of CNCT19 in adult patients with relapsed or refractory acute lymphoblastic leukemia. The study will have the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation & Lymphodepleting Chemotherapy), Treatment and Follow-up, and Survival Follow-up. The total duration of the study is 2 years from CNCT19 cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent is signed by the subject.
2. Age 18 to 65.
3. Relapsed or refractory ALL

   1. Relapse within 12 months of first remission;
   2. Without remission after more than 6 weeks of induction chemotherapy or without remission after 2 cycles of induction chemotherapy regimen;
   3. 2nd or greater Bone Marrow (BM) relapse OR;
   4. First relapse after chemotherapy, without remission after at least 1 rescue treatment;
   5. Any BM relapse after autologous stem cell transplantation (SCT).
4. Documentation of CD19 tumor expression demonstrated in bone marrow or peripheral blood within 3 months of study entry.
5. Patients with Philadelphia chromosome positive (Ph+) ALL are eligible if they are intolerant to or have failed 1 generation and/or 2 generation of tyrosine kinase inhibitor therapy (TKI); no TKI salvage treatments if the patient has a T315I mutation.
6. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening.
7. Eastern cooperative oncology group (ECOG) performance status of 0 to 1.
8. Adequate organ function defined as:

   1. aspartate aminotransferase (AST) ≤ 3 upper limit of normal (ULN);
   2. Serum alanine aminotransferase (ALT) ≤ 3 upper limit of normal (ULN);
   3. Total bilirubin ≤ 2 ULN, except in individuals with Gilbert's syndrome; Note: Patients with Gilbert's syndrome that bilirubin ≤ 3 ULN and direct bilirubin ≤ 1.5 ULN will be eligible;
   4. A serum creatinine≤ 1.5 ULN or Creatine removal rate ≥ 60mL/min (Cockcroft and Gault);
   5. Must have a minimum level of pulmonary reserve as ≤ Grade 1 dyspnea and oxygen saturation > 91% on room air;
   6. International normalized ratio (INR) ≤ 1.5 ULN and activated partial thromboplastin time (APTT) ≤ 1.5 ULN.
9. Have appropriate vascular conditions for apheresis.
10. Non-hematological toxic reactions (excluding diseases related) caused by previous treatment were restored to ≤ 1 level before screening (excluding ≤ 2 level of neurotoxicity caused by hair loss and chemotherapy drugs).
11. Women of childbearing age have a negative blood / urine pregnancy test within 7 days before the CNCT19 infusion. Women of child-bearing potential and all male participants must use highly effective methods of contraception throughout the study and for a period of at least six months after the CNCT19 infusion.

Exclusion Criteria:

1. Active CNS involvement by malignancy.
2. Isolated extra-medullary disease relapse.
3. Patients who received chemotherapy within 2 weeks before CNCT19 infusion. The following situations are excluded:

   1. Lymphodepleting Chemotherapy prescribed by the protocol;
   2. Tyrosine kinase inhibitors (TKI) and hydroxyurea must be stopped > 72 hours prior to CNCT19 infusion;
   3. The following drugs must be stopped > 1 week prior to CNCT19 infusion: 6-mercaptopurine, 6-thioguanine, methotrexate (<25 mg / m2), cytosine arabinoside (<100 mg / m2 / d), vincristine, asparaginase;
   4. Pegylated-asparaginase must be stopped > 4 weeks prior to CNCT19 infusion;
   5. CNS prophylaxis treatment must be stopped > 1 week prior to CNCT19 infusion.
4. Radiotherapy before CNCT19 infusion:

   Non-CNS site of radiation completed < 2 weeks prior to CNCT19 infusion; CNS directed radiation completed < 8 weeks prior to CNCT19 infusion.
5. Therapeutic systemic doses of steroids were stopped < 72 hours prior to CNCT19 infusion. However, the following physiological replacement doses of steroids are allowed: < 10 mg/day hydrocortisone or equivalent.
6. Has had treatment with any prior CAR-T therapy.
7. Patients who have previously received allogeneic hematopoietic stem cell transplantation (allo-HSCT).
8. Patients with systemic vasculitis (such as Wegener granulomatosis, nodular polyarteritis, systemic lupus erythematosus) and active or uncontrolled autoimmune disease (such as autoimmune hemolytic anemia, etc.).
9. Patients who are positive for any of HBsAg, HBeAg, HBeAb, HBcAb, HCV-Ab, TP-Ab.
10. Active malignancy. Patients with Prior malignancy that has been cured for ≥ 2 years are excluded.
11. a. Left Ventricular Ejection Fraction (LVEF) ≤45%; b. III/IV congestive heart failure (NYHA); c. Severe arrhythmia ; QTc≥450ms (male)or QTc≥470ms (female)(QTcB=QT/RR1/2); d.Uncontrolled hypertension (systolic blood pressure ≥140 mmHg and / or diastolic blood pressure ≥90 mmHg) or pulmonary hypertension or unstable angina; e. Myocardial infarction or Coronary Artery Bypass Graft Surgery, heart stent surgery < 6 months prior to CNCT19 infusion; f. Clinically significant valvular disease; g. Other heart diseases that have been judged by the investigator to be unsuitable for receiving cell therapy.
12. Clinically significant pleural effusion.
13. Patients with a history of epilepsy, cerebrovascular ischemia / hemorrhage, cerebellar disease or other active central nervous system diseases.
14. History of deep vein thrombosis or pulmonary embolism within 6 months of screening.
15. Known history of hypersensitivity to ingredients used in the drug.
16. Has had treat with live vaccine within 6 weeks prior to screening.
17. Patients with evidence of currently uncontrollable serious active infections (e.g., sepsis, bacteremia, fungemia, viremia, etc.).
18. Life expectancy < 3 months.
19. Patient in other interventional clinical studies within 3 months before screening, who have received active drug therapy, or who intend to participate in another clinical trial or receive anti-tumor therapy outside the protocol during the entire study.
20. Patients with other conditions making the patients unsuitable for receiving cell therapy as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD), Dose Limiting Toxicity (DLT) and Recommended Phase II Dose (RP2D) | 28 days
  Determine the MTD and DLT of CNCT19 in the Treatment and recommend the dose for Phase II study.
Safety of CNCT19 therapy | 24 months
  Safety measures include adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Overall Remission Rate (ORR), which includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi) | 3 months
  Efficacy of CNCT19 as measured by ORR during the 3 months after CNCT19 infusion, which includes CR and CRi.
Overall Remission Rate (ORR) | 28 days
  Description: ORR includes CR and CRi.
Overall Remission Rate (ORR) with minimal residual disease (MRD) negative bone marrow | 28 days
  MRD negative status as determined by central laboratory using multi-parameter flow cytometry.
Overall Remission Rate (ORR) with minimal residual disease (MRD) negative bone marrow | 3 months
  MRD negative status as determined by central laboratory using multi-parameter flow cytometry.
Overall Remission Rate (ORR) | 6 months
  ORR includes CR and CRi.
Overall Remission Rate (ORR) with minimal residual disease (MRD) negative bone marrow | 6 months
  MRD negative status as determined by central laboratory using multi-parameter flow cytometry.
Duration of remission (DOR) | 24 months
  DOR is defined as the time from the first documented CR or Partial Remission (PR) to the date of the first documented progressive disease(PD) or death due to any cause.
Relapse-free survival (RFS) | 24 Months
  RFS is defined as the time from the documented CR or PR after the CNCT19 infusion to the date of the documented PD or death due to any cause.
Overall survival (OS) | 24 months
  OS is defined as the time from the signing of informed consent form to the date of the last survival follow-up or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Institute of Hematology & Blood Diseases Hospital, Tianjin